CLINICAL TRIAL: NCT00909285
Title: Testing the Effects of TMS Stimulation and Cognitive Training for Alzheimer Patients: A Pilot Study
Brief Title: Effects of Transcranial Magnetic Stimulation (TMS) and Cognitive Training for Alzheimer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Shai Efrati, Assaf Harofeh Medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRX -NC-01
Record Dates: First submitted 2009-05-24; First posted 2009-05-27 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer; TMS; cognitive training
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (#1) (Experimental)
  Interventions: Device: TMS stimulation; Behavioral: Cognitive training
- Control group (#2) (Sham Comparator)
  Interventions: Device: Sham comparator

INTERVENTIONS:
Device: TMS stimulation — TMS stimulation and cognitive training
  Arms: Treatment Group (#1)
Device: Sham comparator — Sham comparator
  Arms: Control group (#2)
Behavioral: Cognitive training — TMS stimulation and cognitive training
  Arms: Treatment Group (#1)

SUMMARY:
Current diagnosis of Alzheimer disease is made by clinical, neuropsychological, and neuroimaging assessments. Routine structural neuroimaging evaluation is based on nonspecific features, such as atrophy, which is a late feature in the progression of the disease. Therefore, developing new approaches for early and specific recognition of Alzheimer disease at the prodromal stages is of crucial importance.

In the present study the investigators would like to examine if combined treatment with TMS and cognitive training (CoTra) for several weeks can produce a sustained improvement in cognitive and behavioral symptomatology of Alzheimer's disease (AD) patients. A number of in vivo neuroimaging techniques, which can be used to reliably and noninvasively assess aspects of neuroanatomy, chemistry, physiology, and pathology, hold promise.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 55-85 years
* Patients diagnosed with early or moderate stage of Alzheimer's disease, according to the DSM-IV criteria.
* MMSE score 15 to 26
* Global Dementia rating 1 or 2
* Physically acceptable for the study as confirmed by medical history and exam, clinical laboratory results and EKG
* Spouse, family member or professional caregiver agree and capable of taking care and responsibility for the participation of the patient in the study (transportation for the patient to and from the investigator's clinic, answering questions regarding the patient's condition and assuming responsibility for medication)
* Written informed consent by patient or legally responsible caregiver.
* Able to undergo MRI scanning sessions (e.g., prior to the onset of the study, upon the attainment of the primary end-point and at the end of the study).
* Commitment to participation in six-to eighteen weeks of the trial regimen consisting of approximately1 hour TMS stimulation and cognitive training daily treatment of five days a week - six to eighteen weeks (and up to two treatments a day in case the Third TMS stimulation and cognitive training Treatment protocol if necessary).

Exclusion Criteria:

* Severe agitation;
* Mental retardation;
* Unstable medical condition;
* Use of benzodiazepines or other hypnotics during the study and preceding two weeks;
* Pharmacological immunosuppression;
* Participation in a clinical trial with any investigational agent within two weeks prior to study enrollment;
* Alcoholism;
* History of Epileptic Seizures or Epilepsy;
* Contraindication for performing MRI scanning;
* Clinically significant abnormal laboratory findings which have not been approved by the Project Director;

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of the TMS stimulation with cognitive training in treatment of early- to mid- stage Alzheimer's patients will be established by improvement of at least 4 points on ADAS-COG. | 3 months

SECONDARY OUTCOMES:
Safety will be established by paucity of related adverse events. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator — Assaf-Harofeh MC
Locations (1):
- Assaf-Harofeh MC, Beer-Yaakov, Israel